CLINICAL TRIAL: NCT03054194
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2730
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2730
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2730-A001-001
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy Participants
Keywords: Healthy participants; E2730; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Dose 1 E2730 (Experimental): Participants will receive Dose 1 of oral E2730 on Day 1.
  Interventions: Drug: E2730
- Cohort 1: Matching placebo (Placebo Comparator): Participants will receive matching oral placebo on Day 1.
  Interventions: Drug: Placebo
- Cohort 2: Dose 2 E2730 (Experimental): Participants will receive Dose 2 of oral E2730 on Day 1.
  Interventions: Drug: E2730
- Cohort 2: Matching placebo (Placebo Comparator): Participants will receive oral matching placebo on Day 1.
  Interventions: Drug: Placebo
- Cohort 3: Dose 3 E2730 (Experimental): Participants will receive Dose 3 of oral E2730 on Day 1.
  Interventions: Drug: E2730
- Cohort 3: Matching placebo (Placebo Comparator): Participants will receive oral matching placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2730 — capsules
  Arms: Cohort 1: Dose 1 E2730; Cohort 2: Dose 2 E2730; Cohort 3: Dose 3 E2730
Drug: Placebo — capsules
  Arms: Cohort 1: Matching placebo; Cohort 2: Matching placebo; Cohort 3: Matching placebo

SUMMARY:
Study E2730-A001-001 is a first-in-human, sequential ascending single dose, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single oral dose of E2730 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, male or female, age ≥18 years and ≤55 years old at the time of informed consent (note: to be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing)
* Body mass index (BMI) ≥18 and <32 kilograms per meters squared (kg/m^2) at Screening

Exclusion Criteria:

* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
* Females who are breastfeeding or pregnant at Screening or Baseline (documented by a negative beta human chorionic gonadotropin [β-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of β-hCG [or hCG]). A negative urine pregnancy test is required before the administration of the first dose per cohort.
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double barrier method [such as condom plus diaphragm with spermicide] or have a vasectomized partner with confirmed azoospermia but hormonal contraceptives are not permitted) throughout the entire study period and for 28 days after study drug discontinuation
  * Are currently abstinent, and do not agree to use a double barrier method (as described above) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation

NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).

* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 3 months after study drug discontinuation.
* Evidence of disease that may influence the outcome of the study within 4 weeks before dosing (eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism)
* Any history of seizures, including those experienced in childhood
* Any history of gastrointestinal surgery that may affect pharmacokinetic profiles of E2730 (eg, hepatectomy, nephrectomy, digestive organ resection) at Screening
* Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening or Baseline
* A prolonged QT/QT corrected (QTc) interval (QC interval corrected using Fridericia's formula [QTcF] >450 milliseconds) demonstrated on ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
* Left bundle branch block at Screening or Baseline
* Persistent systolic blood pressure (BP) >130 or <100 millimeters of mercury (mmHg) or diastolic BP >85 or <50 mmHg at Screening or Baseline
* Persistent heart rate less than 50 beats/min or more than 100 beats/min at Screening or Baseline
* History of myocardial infarction, ischemic heart disease, or cardiac failure at Screening
* History of clinically significant arrhythmia or uncontrolled arrhythmia
* Known history of clinically significant drug allergy at Screening or Baseline
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
* Known to be human immunodeficiency virus positive at Screening
* Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive drug test (including cannabinoids) or alcohol test at Screening or Baseline
* Intake of caffeinated beverages or food within 72 hours before dosing
* Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug-metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussel's sprouts, mustard], and charbroiled meats) within 1 week before dosing
* Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
* Use of prescription drugs within 4 weeks before dosing
* Intake of over-the-counter (OTC) medications within 2 weeks before dosing
* Currently enrolled in another clinical study or used any investigational drug or device within 30 days or 5 half-lives, whichever is longer, preceding informed consent
* Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
* Engagement in strenuous exercise within 2 weeks before check-in (eg, marathon runners, weight lifters)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with any serious adverse event and number of participants with any non-serious adverse event | up to Day 10 (Follow-up/Early Termination)
  An adverse event is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A serious adverse event is defined as any adverse event occurring at any dose that results in any of the following outcomes: results in death; is life threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life function; results in a congenital anomaly/birth defect; or can be defined as any other important medical event.
Number of participants with an abnormal, clinically significant hematology parameter value | Screening; Baseline; Days 2 and 5; Day 10 (Follow-up/Early Termination)
  Participants will fast for at least 4 hours before blood is drawn for the assessment of hematocrit, hemoglobin, platelets, red blood cell (RBC) count, and white blood cell (WBC) count with differential (basophils, eosinophils, lymphocytes, monocytes, neutrophils). Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant blood chemistry parameter value | Screening; Baseline; Days 2 and 5; Day 10 (Follow-up/Early Termination)
  Participants will fast for at least 4 hours before blood is drawn for the assessment of electrolytes (chloride, potassium, sodium); liver function test parameters (alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transpeptidase, direct bilirubin, total bilirubin); renal function test parameters (blood urea/blood urea nitrogen, creatinine); and other parameters such as albumin, calcium, cholesterol, globulin, glucose, lactate dehydrogenase, phosphorus, total protein, triglycerides, and uric acid. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant urine value | Screening; Baseline; Days 2 and 5; Day 10 (Follow-up/Early Termination)
  Urinalysis will be performed to determine abnormalities in the presence of bacteria, casts, crystals, epithelial cells, glucose, ketones, occult blood, pH, protein, RBCs, specific gravity, and WBCs in urine. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant vital sign value | up to Day 10 (Follow-up/Early Termination)
  Vital sign measurements (ie, systolic and diastolic blood pressure [BP] [millimeters of mercury (mmHg)], pulse [beats per minute], respiratory rate [breaths per minute], and body temperature [centigrade]) will be obtained in the supine position by a validated method. Clinical significance will be determined by the Investigator.
Mean change from Baseline in weight | Screening; Baseline; Day 10 (Follow-up/Early Termination)
  Weight (kilograms [kg]) will be obtained by a validated method.
Number of participants with an abnormal, clinically significant electrocardiogram (ECG) parameter value | Screening; Baseline; up to Day 10 (Follow-up/Early Termination)
  An ECG is a record or display of a person's heartbeat produced by electrocardiography. The Holter device will be used for ECG recording. Monitoring will begin at 24 hours before dosing. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant physical examination parameter value | Screening; Baseline; Day 5; Day 10 (Follow-up/Early Termination)
  A comprehensive physical examination will include evaluations of the head, eyes, ears, nose, throat, neck, chest (including heart and lungs), abdomen, limbs, skin, and a complete neurological examination. A urogenital examination will only be required in the presence of clinical symptoms related to those regions. For abbreviated physical examinations, health status will be assessed by brief evaluation of the chest (including heart and lungs), abdomen and limbs, and other physical conditions of note. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant neurological parameter value | Screening
  Abnormalities in neurological parameters due to an increase in inhibitory neurotransmission after E2730 administration will be assessed. Clinical significance will be determined by the Investigator.
Mean maximum observed concentration (Cmax) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  Cmax is defined as the maximum observed concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine Cmax.
Mean time at which the highest drug concentration (tmax) occurs for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  Tmax is defined as the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine tmax.
Mean area under the concentration-time curve from zero time to 24 hours after dosing (AUC[0-24h]) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  AUC represents the total drug exposure over a defined period of time. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine AUC(0-24h).
Mean area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  AUC represents the total drug exposure over a defined period of time. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine AUC(0-t).
Mean area under the concentration-time curve from zero time to 72 hours after dosing (AUC[0-72h]) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  AUC represents the total drug exposure over a defined period of time. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine AUC(0-72h).
Mean area under the concentration-time curve from zero time to 96 hours after dosing (AUC[0-96h]) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  AUC represents the total drug exposure over a defined period of time. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine AUC(0-96h).
Mean area under the concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  AUC represents the total drug exposure over a defined period of time. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine AUC(0-inf).
Mean terminal phase half-life (t1/2) for E2730 and the N-acetyl metabolite in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  Terminal half-life is the time it takes for a substance to lose half of its pharmacological, physiological, or radiologic activity. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine t1/2.
Mean apparent total clearance following extravascular (eg, oral) administration of E2730 (CL/F) in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  CL/F is the rate and extent of absorption and clearance of E2730 from the plasma. Blood samples for the determination of E2730 plasma concentrations will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 will be analyzed to determine CL/F. CL/F will be expressed in volume per time.
Mean apparent volume of distribution at terminal phase (Vz/F) for E2730 in plasma | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  Volume of distribution is defined as the fluid volume that would be required to contain the amount of E2730 present in the body at the same concentration as in the plasma. Vz/F is the apparent volume of distribution at terminal phase for E2730 only. Blood samples for the determination of E2730 plasma concentrations will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 will be analyzed to determine Vz/F.
Metabolite ratio (%) calculated as the ratio of plasma AUC(0-inf) of metabolite to parent following molar correction (MRP) for E2730 and the N-acetyl metabolite | Day 1: predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose. 24 (Day 2), 36 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 216 hours (Day 10) postdose.
  Metabolite ratio (%) is calculated as the ratio of plasma AUC(0-inf) of a metabolite to a parent following molar correction. Blood samples for the determination of E2730 plasma concentrations and its N-acetyl metabolite will be collected from predose through Day 10 (216 hours postdose). Using non-compartmental analysis, plasma concentrations of E2730 and the N-acetyl metabolite will be analyzed to determine the metabolite ratio.

SECONDARY OUTCOMES:
Mean change from Baseline in blood pressure (BP) using ambulatory BP monitoring (ABPM) | Baseline; Day 1; Day 2
  Blood pressure will be measured after the participant has been supine for 10 minutes. At Baseline and at subsequent time points through 24 hours postdose, after supine measurements are completed, participants will be asked to stand up for 2 minutes and BP will then be measured in the standing position. All BP measurements should be performed on the same arm, preferably by the same person. Continuous Mean change from Baseline is calculated as the post-Baseline visit value minus the Baseline value.
Mean change from Baseline in heart rate using Holter monitoring | Baseline; Day 1; Day 2
  Heart rate will be measured after the participant has been supine for 10 minutes. At Baseline and at subsequent time points through 24 hours postdose, after supine measurements are completed, participants will be asked to stand up for 2 minutes and heart rate will then be measured in the standing position. Mean change from Baseline is calculated as the post-Baseline visit value minus the Baseline value.
Mean change from Baseline in corrected QT (QTc) interval using Holter monitoring | Baseline; Day 1; Day 2
  ECGs will be extracted from the Holter device on Day 1 at predose and postdose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, and 12 hours; and on Day -1 at times matching those on Day 1 (from 24 hours predose on Day -1 until predose on Day 1). On Day 2 (24 hours postdose), ECGs will again be extracted from the Holter device (24 hours postdose). High-precision QT analyses (HPQT) will be performed using data extracted from the 24-hour Holter recording. QT interval corrected for heart rate using Friderica's formula (QTcF) intervals will be estimated and used for the HPQT analyses. Other correction methods such as QTc (individual) and QT beat-to-beat (QTbTb) may be used if QTcF is not deemed to be appropriate. Mean change from Baseline is calculated as the post-Baseline visit value minus the Baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No